CLINICAL TRIAL: NCT03101800
Title: Low-dose Azathioprine and Allopurinol- Versus Azathioprine Monotherapy in Patients With Ulcerative Colitis: An Investigator-initiated, Open, Multicentre, Parallel-arm, Randomised Controlled Trial
Brief Title: Beneficial and Harmful Effects of Azathioprine and Allopurinol Versus Standard Azathioprine Therapy for Patients With Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Zealand University Hospital (Other); University of Copenhagen (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Viborg Regional Hospital (Other); Vejle Hospital (Other); Sydvestjysk Hospital Esbjerg (Unknown)
Responsible Party: Principal Investigator, Sandra Bohn Thomsen, MD, Ph.D. candidate, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAUC Study
Record Dates: First submitted 2017-01-27; First posted 2017-04-05 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Colitis, Ulcerative; Colitis Ulcerative Exacerbation
Keywords: Azathioprine; Allopurinol; Antimetabolites; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Azathioprine; Allopurinol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azathioprine and Allopurinol (Experimental)
  Interventions: Drug: Azathioprine and Allopurinol
- Azathioprine (Active Comparator)
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Azathioprine and Allopurinol — Low dose Azathioprine in combination with allopurinol 100 mg for 1 year
  Arms: Azathioprine and Allopurinol
Drug: Azathioprine — Standard weight based azathioprine dosage
  Arms: Azathioprine

SUMMARY:
Azathioprine is considered first line immunomodulatory therapy for patients with ulcerative colitis. Up to 50% are treatment failures or experience adverse events leading to treatment withdrawal. Recent evidence suggests that the combination of allopurinol and low dose azathioprine increases the proportion of treatment responders and reduce the risk of adverse events.

Objectives: To evaluate the beneficial and harmful effects of low dose azathioprine and allopurinol versus standard azathioprine monotherapy in patients with ulcerative colitis.

DETAILED DESCRIPTION:
Investigator initiated, multicentre, parallel arm, open, randomised controlled trial with blinded assessment

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all trial procedures and being available for the duration of the trial.
* Clinically and histologically verified ulcerative colitis eligible for treatment with thiopurines due to steroid dependence (failure to taper steroid or starting a second course of systemic steroids within 1 year) or patients with the need for rescue therapy with anti-TumorNecrosisFactorα (anti-TNFα)
* A sigmoidoscopy or colonoscopy showing active inflammation during the present disease flare
* Negative stool test for pathogen bacteria incl. Clostridium difficile
* Informed consent.
* Normal TPMT genotype (homozygous wild-type).
* Oral 5-Asa dose stable for 2 weeks

Exclusion Criteria:

* Kidney disease with a GlomerularFiltration Rate (GFR) < 50 ml/min.
* Persistent alanine aminotransferase U/L (ALT) twice above upper limit of the normal range.
* Participation in other interventional clinical trials.
* Pregnancy or breastfeeding.
* Previous thiopurin treatment.
* Previous or current treatment with other biologics than anti-TNFα
* Not being able to comply with the study, assessed by investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-12-14 (Actual); Primary Completion 2019-11-14 (Estimated); Study Completion 2019-12-14 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 52 weeks
  Steroid- and biologic treatment free remission defined as total Mayo score ≤1 without rectal bleeding.

SECONDARY OUTCOMES:
Time to remission | 52 weeks
Clinical response | 52 weeks
  defined as a Mayo score between ≤1 to < 3
Endoscopic remission | 52 weeks
  defined as a Mayo subscore of 0
Fecal calprotectin | 52 weeks
Histological mucosal healing | 52 weeks
Quality of life (SIBDQ) | 52 weeks
  Using Inflammatory Bowel Disease Questionnaire Quality of life (SIBDQ)
Quality of life (SHS) | 52 weeks
  Using the Short health scale (SHS)
Correlation between 6ThioGuanineNucleotiude (6TGN) and clinical mayo score | From week 6 to week 52
Correlation between 6TGN and standard blood tests | From week 6 to week 52
Correlation between 6TGN and fecal calprotectin | From week 6 to week 52
Correlation between 6TGN endoscopic mayo score | From week 6 to week 52
Correlation between 6TGN and histological mucosal healing | From week 6 to week 52
Adverse events | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre university hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523
- [Derived] Kiszka-Kanowitz M, Theede K, Thomsen SB, Bjerrum JT, Brynskov J, Gottschalck IB, Akimenko E, Hilsted KL, Neumann A, Wildt S, Larsen L, Munk JK, Ibsen PH, Janjua HGR, Gluud LL, Mertz-Nielsen A. Low-dose azathioprine and allopurinol versus azathioprine monotherapy in patients with ulcerative colitis (AAUC): An investigator-initiated, open, multicenter, parallel-arm, randomised controlled trial. EClinicalMedicine. 2022 Mar 5;45:101332. doi: 10.1016/j.eclinm.2022.101332. eCollection 2022 Mar. PMID 35274092